CLINICAL TRIAL: NCT04947956
Title: Camrelizumab in Patients With Unresectable Hepatocellular Carcinoma in China: a Real-world Study
Brief Title: Camrelizumab in Patients With Unresectable Hepatocellular Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Principal Investigator, Jian Zhou, Chief physician, Shanghai Zhongshan Hospital
Other Study IDs: MA-HCC-RWS-008
Record Dates: First submitted 2021-06-29; First posted 2021-07-01 (Actual); Last update posted 2021-07-01 (Actual); Status verified 2021-06

CONDITIONS: Unresectable Hepatocellular Carcinoma
MeSH Terms: interventions — camrelizumab; apatinib; Radiotherapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Camrelizumab — The camrelizumab-based treatment will be determined by the investigator.
  Other Names: Apatinib, TACE, Radiotherapy, et al

SUMMARY:
Primary liver cancer is the second most common cause of cancer death in China, and hepatocellular carcinoma (HCC) represents more than 80% of liver cancer cases. The majority of HCC cases present at an advanced stage, and are thus not amenable to surgery. Immunotherapies, including PD-1 and PD-L1 inhibitors, alone or combined with other regimens, have shown encouraging clinical activity in unresectable HCC. Camrelizumab, a humanised monoclonal antibody against PD-1, has been shown to block the binding of PD-1 to PD-L1 and consequently inhibit the immune escape of tumour cells， which has been approved for the second-line treatment of advanced HCC. This observational study aims to evaluate the safety and efficacy of camrelizumab in Chinese unresectable HCC in the real world.

DETAILED DESCRIPTION:
Primary liver cancer is the second most common cause of cancer death in China, and hepatocellular carcinoma (HCC) represents more than 80% of liver cancer cases. The majority of HCC cases present at an advanced stage, and are thus not amenable to surgery. Immunotherapies, including PD-1 and PD-L1 inhibitors, alone or combined with other regimens, have shown encouraging clinical activity in unresectable HCC. Camrelizumab, a humanised monoclonal antibody against PD-1, has been shown to block the binding of PD-1 to PD-L1 and consequently inhibit the immune escape of tumour cells，which has been approved for the second-line treatment of advanced HCC. This multi-center, open-label, observational study aims to evaluate the safety and efficacy of camrelizumab in Chinese unresectable HCC in the real world. This study also aims to evaluate the treatment of camrelizumab in subgroups, to provide information of treatment regimens and efficacy in clinical practice. The anticipated sample size is 1000, and the camrelizumab-based treatment will be determined by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* 1. Volunteer to participate in this study and sign an informed consent form; 2. Age ≥ 18 years; 3. Hepatocellular carcinoma confirmed/clinically confirmed by histopathology, cytology or imaging

Exclusion Criteria:

* 1. Documented pregnant or breastfeeding women;
* 2. Patients who are participating in any interventional trials beyond clinical practice.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Unresectable hepatocellular carcinoma
Sampling Method: Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2023-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
The incidence of treatment-emergent adverse events (TEAE) | Up to ~2 years
  The incidence of treatment-emergent adverse events (TEAE)

SECONDARY OUTCOMES:
Overall survival | Up to ~2 years
  Overall survival
Progression-free survival | Up to ~2 years
  Progression-free survival
Time to progression | Up to ~2 years
  Time to progression

REFERENCES:
- [Background] Qin S, Ren Z, Meng Z, Chen Z, Chai X, Xiong J, Bai Y, Yang L, Zhu H, Fang W, Lin X, Chen X, Li E, Wang L, Chen C, Zou J. Camrelizumab in patients with previously treated advanced hepatocellular carcinoma: a multicentre, open-label, parallel-group, randomised, phase 2 trial. Lancet Oncol. 2020 Apr;21(4):571-580. doi: 10.1016/S1470-2045(20)30011-5. Epub 2020 Feb 26. PMID 32112738
- [Background] Bray F, Ferlay J, Soerjomataram I, Siegel RL, Torre LA, Jemal A. Global cancer statistics 2018: GLOBOCAN estimates of incidence and mortality worldwide for 36 cancers in 185 countries. CA Cancer J Clin. 2018 Nov;68(6):394-424. doi: 10.3322/caac.21492. Epub 2018 Sep 12. PMID 30207593
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Mo H, Huang J, Xu J, Chen X, Wu D, Qu D, Wang X, Lan B, Wang X, Xu J, Zhang H, Chi Y, Yang Q, Xu B. Safety, anti-tumour activity, and pharmacokinetics of fixed-dose SHR-1210, an anti-PD-1 antibody in advanced solid tumours: a dose-escalation, phase 1 study. Br J Cancer. 2018 Aug;119(5):538-545. doi: 10.1038/s41416-018-0100-3. Epub 2018 May 14. PMID 29755117
- [Background] Huang J, Xu B, Mo H, Zhang W, Chen X, Wu D, Qu D, Wang X, Lan B, Yang B, Wang P, Zhang H, Yang Q, Jiao Y. Safety, Activity, and Biomarkers of SHR-1210, an Anti-PD-1 Antibody, for Patients with Advanced Esophageal Carcinoma. Clin Cancer Res. 2018 Mar 15;24(6):1296-1304. doi: 10.1158/1078-0432.CCR-17-2439. Epub 2018 Jan 22. PMID 29358502
- [Background] Xu J, Shen J, Gu S, Zhang Y, Wu L, Wu J, Shao G, Zhang Y, Xu L, Yin T, Liu J, Ren Z, Xiong J, Mao X, Zhang L, Yang J, Li L, Chen X, Wang Z, Gu K, Chen X, Pan Z, Ma K, Zhou X, Yu Z, Li E, Yin G, Zhang X, Wang S, Wang Q. Camrelizumab in Combination with Apatinib in Patients with Advanced Hepatocellular Carcinoma (RESCUE): A Nonrandomized, Open-label, Phase II Trial. Clin Cancer Res. 2021 Feb 15;27(4):1003-1011. doi: 10.1158/1078-0432.CCR-20-2571. Epub 2020 Oct 21. PMID 33087333